CLINICAL TRIAL: NCT01442714
Title: Azacitidine Plus Lenalidomide Combination in Elderly Patients With Previously Treated Acute Myeloid Leukemia (AML) & High-Risk Myelodysplastic Syndromes (MDS) (VIREL2 Trial)
Brief Title: Azacitidine + Lenalidomide Combo in the Elderly With Previously Treated AML & High-Risk MDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy - Inability to meet the primary response endpoint
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Bruno C. Medeiros, Associate Professor Medicine Hematology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21686; SU-08122011-8268 (Other: Stanford University); HEM0022 (Other: OnCore Number); VIREL2 (Other: Stanford University)
Record Dates: First submitted 2011-09-23; First posted 2011-09-28 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Leukemia; Acute Myeloid Leukemia (AML); Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine plus Lenalidomide (Experimental): Patients will receive a single dose of azacitidine 75 mg/m² SC or IV on days 1 to 7, followed by lenalidomide 50 mg PO daily on days 8 to 28 of a 42-day cycle.
  Interventions: Drug: Azacitidine; Drug: Lenalidomide

INTERVENTIONS:
Drug: Azacitidine — Azacitidine is a chemical analogue of the cytosine nucleoside used in DNA and RNA. Azacitidine is thought to induce antineoplastic activity via two mechanisms; inhibition of DNA methyltransferase at low doses, causing hypomethylation of DNA, and direct cytotoxicity in abnormal hematopoietic cells in the bone marrow through its incorporation into DNA and RNA at high doses, resulting in cell death
  Other Names: 5-azacytidine; Vidaza
Drug: Lenalidomide — Lenalidomide has been used to successfully treat both inflammatory disorders and cancers. In vitro, lenalidomide has three main activities: direct anti-tumor effect, inhibition of angiogenesis, and immunomodulatory role. In vivo, lenalidomide induces tumor cell apoptosis directly and indirectly by inhibition of bone marrow stromal cell support, by anti-angiogenic and anti-osteoclastogenic effects, and by immunomodulatory activity.
  Other Names: CC-5013; Celgene; Revlimid

SUMMARY:
The purpose of the trial is to study how the elderly patients who have previously undergone treatment for acute myeloid leukemia and high-rRisk myelodysplastic syndromes, respond to a combined treatment with azacitidine and lenalidomide.

DETAILED DESCRIPTION:
This is an open label, single-center, and phase 2 study of the combination of azacitidine with lenalidomide in previously treated elderly patients with acute myeloid leukemia (AML) and/or high-risk myelodysplastic syndrome (MDS) who have failed prior therapy with either a demethylating agent and/or IMIDs. MDS includes Chronic Myeloid Leukemia (CML).

Participants patients will receive azacitidine on the first 7 days followed by lenalidomide. Disease assessments with bone marrow examinations will be performed and if a complete response (CR); Complete remission with incomplete count recovery (CRi); partial response (PR); or stable disease (SD) is documented after 6 total cycles, participants will continue treatment until evidence of disease progression, provided they are tolerating treatment. Participants who have progressive disease or relapsed disease after the 6th cycle will be taken off the study, and participants with excessive toxicity at any time will be taken off the study.

* CR = Less than 5% blasts with no Auer rods, absence of extramedullary disease, absolute neutrophil count (ANC) > 1000/µL, platelets > 100,000/µL, and independence of red cell transfusion)
* CR with incomplete recovery (CRi) = all criteria of a CR with the exception of a platelet count less than 100,000/µL or residual neutropenia (< 1000/µL).
* PR = Meeting all hematologic criteria for CR with an allowance for 5% to 25% bone marrow blasts or decrease of pretreatment bone marrow blast percentage by ≥ 50%.
* SD = Change in bone marrow aspirate blast count within 10% of baseline.
* PD = Progressive / relapsed disease defined as reappearance of blasts in the blood or bone marrow blasts ≥ 5%, and development of extramedullary disease.

ELIGIBILITY:
Inclusion Criteria:

* acute myeloid leukemia (AML) (according to the WHO 2008 classification):

  * De novo
  * Secondary AML previously treated with demethylating agents for AML
  * Secondary AML previously treated with demethylating agents for MDS
  * Secondary AML previously treated with high dose lenalidomide for AML (≥ 25mg)
* High Risk MDS:

  * Del (5q)
  * Non-del (5q), previously-treated with lenalidomide.
  * Novo or secondary HR-MDS previously treated with demethylating agents
* White blood cell (WBC) ≤ 10,000
* Age ≥ 60
* Not an immediate candidate for allogeneic stem cell transplantation
* Unwilling or unable to receive conventional chemotherapy
* Prior therapy:

  * with single agent demethylator (5-Azacitidine or Decitabine)
  * with Lenalidomide
* Eastern Cooperative Oncology Group performance status ≤ 2
* Life expectancy > 2 months
* All study participants must be registered into the mandatory RevAssist program
* Willing and able to comply with the requirements of RevAssist
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test 10-14 days prior to study enrollment and again within 24 hours of prescribing lenalidomide

  * Must commit to either continued abstinence from intercourse or begin two acceptable methods of birth control, at least 28 days before she starts taking lenalidomide.
  * Must also agree to ongoing pregnancy testing.
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Willing and able to understand and voluntarily sign a written informed consent
* Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Patients with LR-MDS progressing to HR-MDS after low dose lenalidomide or 5-day azacitidine will not be eligible.
* History of intolerance to thalidomide

  -development of erythema nodosum while taking thalidomide or similar drugs
* Known or suspected hypersensitivity to azacitidine or mannitol
* Patients with advanced malignant hepatic tumors.
* Concomitant treatment with other anti-neoplastic agents, with the exception of hydroxyurea
* Previous participation on the VIREL study with the concomitant use of azacitidine plus lenalidomide.
* Anti-neoplastic treatment less than four weeks prior to enrollment, with the exception of hydroxyurea
* Use of any other experimental drug or therapy within 28 days of baseline
* Inability to swallow or absorb drug
* Active opportunistic infection or treatment for opportunistic infection within four weeks of first day of study drug dosing
* New York Heart Association Class III or IV heart failure
* Unstable angina pectoris
* Uncontrolled cardiac arrhythmia
* Uncontrolled psychiatric illness that would limit compliance with requirements
* Known HIV infection
* Pregnant
* Breast feeding
* Lactating females must agree not to breast feed while taking lenalidomide
* Other medical or psychiatric illness or organ dysfunction or laboratory abnormality
* Laboratory abnormalities:

  * Either creatinine ≥ 1.5 mg / dL or creatinine clearance ≤ 50 mL / min
  * Total bilirubin >1.5 x institutional ULN
  * AST and ALT > 2.5 x institutional ULN

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Carneiro de Medeiros, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Azacitidine Plus Lenalidomide: Patients will receive a single dose of azacitidine 75mg/m2 SC/IV on d 1 to 7, followed by lenalidomide 50mg PO daily on d 8 to 28 of a 42-day cycle.
  Azacitidine is a chemical analogue of the cytosine nucleoside used in DNA and RNA. Azacitidine is thought to induce antineoplastic activity via two mechanisms; inhibition of DNA methyltransferase at low doses, causing hypomethylation of DNA, and direct cytotoxicity in abnormal hematopoietic cells in the bone marrow through its incorporation into DNA and RNA at high doses, resulting in cell death
  Lenalidomide: Lenalidomide has been used to successfully treat both inflammatory disorders and cancers. In vitro, lenalidomide has three main activities: direct anti-tumor effect, inhibition of angiogenesis, and immunomodulatory role. In vivo, lenalidomide induces tumor cell apoptosis directly and indirectly by inhibition of bone marrow stromal cell support, by anti-angiogenic and anti-osteoclastogenic effects, and by immunomodulatory
Period: Overall Study
Arm/Group | Azacitidine Plus Lenalidomide
Started | 33
Completed | 21
Not Completed | 12
Not completed — Death | 11
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Azacitidine Plus Lenalidomide: Azacitidine + Lenalidomide Combo
Arm/Group | Azacitidine Plus Lenalidomide
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS Scale:
  0 Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead
  Participants
    0 | 24
    1 | 6
    2 | 3
    Not eligible | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the sum of Complete Response (CR) + CR with incomplete count recovery (CRi) + Partial Response (PR).
Time Frame: 203 days
Measure: Count of Participants; unit: Participants
Groups:
- Azacitidine Plus Lenalidomide: Acute myeloid leukemia (AML) ORR was defined as the sum of Complete Response (CR) + CR with incomplete count recovery (CRi) + Partial Response (PR): (CR + CRi + PR)
Arm/Group | Azacitidine Plus Lenalidomide
Number analyzed (Participants) | 33
Participants | 5

2. Secondary Outcome: Median Duration of Response
Description: The median duration of response was defined by the median duration of response for participants with Complete Response (CR); CR with incomplete count recovery (CRi); or Partial Response (PR).
Time Frame: 203 days
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Azacitidine Plus Lenalidomide: Patients will receive a single dose of azacitidine 75mg/m2 SC/IV on d 1-7, followed by lenalidomide 50mg PO daily on d 8-28 of a 42-day cycle.
  Azacitidine is a chemical analogue of the cytosine nucleoside used in DNA and RNA. Azacitidine is thought to induce antineoplastic activity via two mechanisms; inhibition of DNA methyltransferase at low doses, causing hypomethylation of DNA, and direct cytotoxicity in abnormal hematopoietic cells in the bone marrow through its incorporation into DNA and RNA at high doses, resulting in cell death. Lenalidomide: Lenalidomide has been used to successfully treat both inflammatory disorders and cancers. In vitro, lenalidomide has three main activities: direct anti-tumor effect, inhibition of angiogenesis, and immunomodulatory role. In vivo, lenalidomide induces tumor cell apoptosis directly and indirectly by inhibition of bone marrow stromal cell support, by anti-angiogenic and anti-osteoclastogenic effects, and by immunomodulatory.
Arm/Group | Azacitidine Plus Lenalidomide
Number analyzed (Participants) | 5
days | 118 [56.48 to 349.5]

3. Secondary Outcome: Overall Survival
Description: Survival was measured from the 1st day of azacitidine treatment to death from any cause.
Time Frame: 462 Days
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine Plus Lenalidomide
Number analyzed (Participants) | 33
months | 5 [3.7 to 8.6]

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | Azacitidine Plus Lenalidomide
All-Cause Mortality (participants affected / at risk) | 30/33
Serious Adverse Events (participants affected / at risk) | 33/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine Plus Lenalidomide (N=33)
Neutropenic fever (Infections and infestations) | 25 — Including: Neutropenia
Respiratory complications (Respiratory, thoracic and mediastinal disorders) | 8 — Including: dyspnea, pneumonia, aspiration pneumonitis
Diarrhea (Gastrointestinal disorders) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Sepsis (Infections and infestations) | 2 — including: sepsis with acute dysfunction
Death on study (Respiratory, thoracic and mediastinal disorders) | 11
Cardiac complications (Cardiac disorders) | 2 — Including: atrial flutters, asystole
Pancytopenia (Blood and lymphatic system disorders) | 2
Colon Volvulus (Gastrointestinal disorders) | 1
Neck pain and stiffness (Musculoskeletal and connective tissue disorders) | 1
Progressive disease (Infections and infestations) | 2 — worsening AML
Cellulitis (General disorders) | 2 — right groin and facial (periorbital)
Generalized weakness (Musculoskeletal and connective tissue disorders) | 2 — lethargic
Graft vs host disease (GvHD) (General disorders) | 1
Neck complications (Infections and infestations) | 2 — Including: abscess, pain and stiffness
Rigors secondary to fever (General disorders) | 1
Body pain (Musculoskeletal and connective tissue disorders) | 2 — back, abdomen
Encephalopathy (Nervous system disorders) | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 — (DIC)
Vomitting (Gastrointestinal disorders) | 1
Skin infections (Skin and subcutaneous tissue disorders) | 2 — sweet syndrome
Hypoxia (Musculoskeletal and connective tissue disorders) | 1
Fever (General disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine Plus Lenalidomide (N=33)
Neuropathy (Nervous system disorders) | 2 — In feet and fingers. Includes Peripheral Neuropathy.
Edema (Musculoskeletal and connective tissue disorders) | 2 (2) — on lower extremities
apneic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Crackles at right base of lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cramps (Musculoskeletal and connective tissue disorders) | 2 (2) — Upper and lower extremities
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Difficulty urinating (Renal and urinary disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fungal pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Left carotid (Cardiac disorders) | 2 (2) — artery stenosis and endarterectomy
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
skin nodules (Skin and subcutaneous tissue disorders) | 2 (2)
Tachycardiac (Cardiac disorders) | 1 (1)
Ecchymoses on site injections (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated LFT (AST>AST) (Renal and urinary disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
erythema and conjunctival injection of right eye (Infections and infestations) | 2 (2) — including hemorrhaging and swelling
erythematous lesions at injection site at abdomen (Infections and infestations) | 1 (1)
Fall (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
fracture of left fibula (General disorders) | 1 (1)
Frontal headache (General disorders) | 1 (1)
Hoarse voice (Respiratory, thoracic and mediastinal disorders) | 3 (3)
hyperglycemic (Blood and lymphatic system disorders) | 1 (1)
Hypotensive (Blood and lymphatic system disorders) | 1 (1)
Hypertrophy of her gums (Blood and lymphatic system disorders) | 1 (1)
epigastic pain after eating (Gastrointestinal disorders) | 1 (1) — intermittent
episodes of chest pressure (Cardiac disorders) | 1 (1) — intermittent
Large bruise (Skin and subcutaneous tissue disorders) | 1 (1) — on right tight
Left hip injury (General disorders) | 1 (1)
Left leg pain (General disorders) | 3 (3) — including sciatica and cramping
left thyroid nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mild erythema at abdominal injection site (General disorders) | 1 (1)
Mouth soures/ thrush (General disorders) | 4 (4) — including oral ulcer
Night sweat (General disorders) | 2 (2)
Nose bleeds (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Open sore of lower lip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Redness and itching of eyes (Eye disorders) | 1 (1)
Tremors (Musculoskeletal and connective tissue disorders) | 2 (2)
Significant Cytopenias (Blood and lymphatic system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sore tongue (Respiratory, thoracic and mediastinal disorders) | 2 (2)
stress incontinence (General disorders) | 1 (1)
Sudden loss of central vision (Eye disorders) | 1 (1)
Swollen Knee (General disorders) | 1 (1)
Taste changes (Respiratory, thoracic and mediastinal disorders) | 1 (1)
tender facial skin (General disorders) | 1 (1)
Unspecified arrhythmia (Cardiac disorders) | 1 (1)
weight loss (General disorders) | 1 (1)
Allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes